CLINICAL TRIAL: NCT07171099
Title: Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Clinical Trial of the Efficacy and Safety of Rengalin in the Treatment of Cough in Acute Viral Upper Respiratory Tract Infections Tract Infections in Children During the Epidemic Growth of Influenza and ARVI
Brief Title: Efficacy and Safety of Rengalin in the Treatment of ARVI Cough in Children
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-RN-008
Record Dates: First submitted 2025-07-14; First posted 2025-09-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-06

CONDITIONS: Cough
Keywords: Cough; Upper respiratory infection; Children from 6 months to 3 years
MeSH Terms: conditions — Cough; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized, parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rengalin (Experimental): Orally. 5 ml per dose 3 times a day for 7 days. The drug is taken without meals.
  Interventions: Drug: Rengalin
- Placebo (Placebo Comparator): Placebo using the dosing regimen Rengalin for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rengalin — Solution for oral administration
  Arms: Rengalin
Drug: Placebo — Solution for oral administration
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of liquid dosage form of Rengalin in the treatment of cough in acute viral upper respiratory tract infections infections in children in during the epidemic growth of influenza and ARVI. The main questions it aims to answer are:

Investigators will compare the liquid dosage form of Rengalin to a placebo (a look-alike substance that contains no drug) to see if Rengalin in the liquid dosage form works for cough in acute viral upper respiratory tract infections in children.

Participants will:

Take the liquid dosage form of Rengalin or placebo per os 5 ml per administration 3 times a day for 7 days.

DETAILED DESCRIPTION:
The design is a multicenter, double-blind, placebo-controlled, randomized, parallel-group clinical trial evaluating the efficacy and safety of the study therapy.

The trial will enroll children of either gender aged 6 months to 3 years, who consulted a physician for dry/non-productive cough caused by acute viral upper respiratory tract infections during the seasonal growth of influenza and ARVI.

The duration of cough at inclusion in the trial should be at least 24 hours but not more than 72 hours; cough severity - 6 or more points (according to the Cough Severity Score (CSS)).

After one of the parents/adoptive parents signs the patient information leaflet (PIL) and the informed consent form (ICF) (two versions are used - with the consent of the parent/adoptive parent to take blood and urine samples for the purpose of conducting laboratory tests or without consent) for participation in the clinical trial at Visit 1, complaints and anamnesis are collected, vital signs are assessed, a physical examination is performed, concomitant therapy is recorded, and laboratory tests are conducted.

It is planned to conduct a general urine analysis, general and biochemical blood tests in at least 50% of patients.

At Visit 1, the physician together with the parent/adoptive parent fills out the CSS scale.

If inclusion criteria are met and there are no any exclusion criteria at Visit 1 (Day 1), the patient is enrolled in the study and randomized to one of two groups: Group 1 patients will receive Rengalin; Group 2 patients will receive Placebo.

After three days of the study therapy, at Visit 2 (Day 4), the physician evaluates the patient's condition and adjusts the therapy. If there are indications (secretion of viscous sputum), the physician prescribes the mucolytic ambroxol; at the same time, patients of group 1 continue taking Rengalin, and patients of group 2 continue taking Placebo.

The study will use an electronic patient diary (EPD) in which the parent/adoptive parent will record the severity of daytime and nighttime cough as measured by the CSS during the 7 days the patient is in the study. In addition, any possible worsening of the patient's condition (if applicable) will be recorded in the EPD for safety assessment and recording of adverse events.The investigator will instruct parents/adoptive parents will instruct parents/adoptive parents on how to fill out the diary.

The parent/adoptive parent will make the first marks on the cough severity scale in the EDS together with the physician at Visit 1. The EPD will be available for completion throughout the patient's participation in the study. Twice a day, the parent/adoptive parent will receive an SMS reminder: "Please mark the severity of daytime and nighttime cough in the diary. Do not forget to take the medication given to you." The patient treatment continues for 7 days, observation - for 14 days (screening, randomization - 1 day, treatment - 7 days, follow-up - up to 14 days; delayed "phone visit" - 14 days).

On days 4 (Visit 2) and 8 (Visit 3), two visits are planned (at home or at a medical center), during which the physician collects complaints, records medical examination data, identifies possible bacterial complications of acute respiratory infections, monitors prescribed and concomitant therapy, evaluates the safety of the treatment, and checks the filling of the CSS in the EPD.

At Visit 3 (Day 8), samples are collected for laboratory testing. The study drug that the parent/adopter received at Visit 1 must be returned at Visit 3 to assess compliance with the study therapy.

If the patient's condition worsens, the doctor make an unscheduled visit. "Telephone visit" (Visit 4, Day 14±1) is conducted to interview parents/adoptive parents about the patient's condition, presence/absence of cough, bacterial complications of acute respiratory viral infections, and the possible use of antibacterial drugs.

During the study, the use of antiviral drugs, symptomatic agents, and drugs for the treatment of concomitant diseases is permitted, with the exception of drugs listed in the section "Prohibited concomitant therapy".

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients of both genders aged over 6 months and under 3 years.
2. Clinically confirmed diagnosis of acute viral upper respiratory tract infections (acute pharyngitis, nasopharyngitis, tonsillitis, laryngitis, laryngotracheitis, tracheitis, acute viral respiratory infection of multiple and unspecified localization) during the epidemic growth of influenza and ARVI.
3. Dry (non-productive) cough lasting at least 24 hours but not more than 72 hours.
4. Total (day and night) cough severity score of 6 or more.
5. Availability of a patient information sheet and an informed consent form for participation in the clinical trial signed by one of the patient's parents/adoptive parents.

Exclusion Criteria:

1. Presence of the following diseases at the time of inclusion in the clinical trial:

   1.1 Inflammatory processes in the lower respiratory tract. 1.2 Grade III adenoid hypertrophy. 1.3 Chronic adenoiditis. 1.4 Postnasal drip syndrome. 1.5 Gastroesophageal reflux. 1.6 Bronchial asthma. 1.7 Cystic fibrosis. 1.8 Primary ciliary dyskinesia 1.9 Bronchopulmonary dysplasia 1.10 Malformations of the respiratory and ENT organs 1.11 Other chronic lung diseases. 1.12 Primary/secondary immunodeficiency. 1.13 Oncological disease of any localization.
2. Suspected bacterial infection of any localization, including pneumonia, sinusitis, otitis media.
3. Allergic rhinitis.
4. Bronchial obstruction syndrome.
5. Acute obstructive laryngitis [croup] and epiglottitis.
6. Congenital heart defects with hypervolemia in pulmonary circulation.
7. Acute respiratory failure.
8. Inflammatory, degenerative, demyelinating diseases of the central nervous system, polyneuropathies, epilepsy.
9. Exacerbation or decompensation of chronic diseases affecting the patient's ability to participate in a clinical trial.
10. Presence of allergy/hypersensitivity to any components of the medicines used in the treatment.
11. Taking medications listed in the section "Prohibited Concomitant Therapy" within 4 weeks prior to inclusion in the study.
12. Patients whose parents/adoptive parents, from the investigator's point of view, will not comply with observation requirements during the study or with the administration of study drugs.
13. Participation in other clinical trials within 3 months prior to inclusion in this trial.
14. A patient's parent/adoptive parent is related to on-site research personnel directly involved in the trial, or is the immediate family member of the investigator. 'Immediate family members' mean spouses, parents, children, or siblings, whether related or adopted.
15. The patient's parent/adoptive parent is employed by OOO "NPF "MATERIA MEDICA HOLDING", i.e., is an employee of the company, a temporary contract employee, or a designated official responsible for conducting the trial or their immediate family member.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients responded to treatment | On baseline and 3 day
  The percentage of patients responded to treatment (reduction in the total (day and night) cough severity score to 3 points or less after 3 days of treatment - isolated cough episodes or complete absence of cough during the day) after 3 days.

SECONDARY OUTCOMES:
Change in the total CSS | On baseline and 7 day
  Change in the total Cough Severity Score (daytime and nighttime) after 7 days of treatment compared to baseline. The minimum value - 0 (no cough) and maximum value - 10 (severe cough).

OTHER OUTCOMES:
Percentage of patients without daytime cough | On baseline and 7 day
  Percentage of patients with no daytime cough acording to Cough Severity Score (SCC) after 7 days of treatment. The minimum value - 0 (no cough) and maximum value - 5 (severe cough).
Percentage of patients with a decrease in daytime cough | On baseline and 7 day
  Percentage of patients with a decrease in daytime cough severity ≤ 1 point on the Cough Severity Score (SCC) after 7 days of treatment. The minimum value - 0 (no cough) and maximum value - 5 (severe cough).
Percentage of patients without night cough | On baseline and 7 day
  Percentage of patients with no night cough (0 points according to the Cough Severity Score (SCC)) after 7 days of treatment. The minimum value - 0 (no cough) and maximum value - 5 (severe cough).
Percentage of patients with a reduction in nighttime cough | On baseline and 7 day
  Percentage of patients with a reduction in nighttime cough severity ≤ 1 point on the Cough Severity Score (SCC) after 7 days of treatment. The minimum value - 0 (no cough) and maximum value - 5 (severe cough).
Cough severity | 7 days
  Cough severity during 7 days of treatment (based on the area under the curve (AUC) of daytime and nighttime cough scores). The area under the curve is determined in conventional units (points multiplied by days).
Percentage of patients prescribed the ambroxol | On 4 day
  Percentage of patients who were additionally prescribed the mucolytic ambroxol on the 4th day of treatment.
Proportion of patients required antibacterial drugs or hospitalization | 14 days of treatment
  Proportion of patients with worsening ARVI course (bacterial complications of ARVI that required antibacterial drugs or hospitalization) within 14 days of participation in the trial.
Number of patients with adverse events (AEs) | From day 1 to day 14
  The presence of adverse events. Based on medical records.
Severity of AEs | From day 1 to day 14
  Number of patients with the intensity (severity) of adverse events. Based on medical records.
Causal relationship of AEs to the sudy drug | From day 1 to day 14
  The causal relationship to the study drug of adverse events. Based on medical records. The assessment of causality is made by the investigator based on his/her clinical opinion (certain, probable, doubtful, conditional, unclassifiable, not related).
Outcome of AEs | From day 1 to day 14
  The outcome of adverse events. Based on medical records. The outcome of AE is made by investigator (recovery/resolution, incomplete recovery/resolution, no recovery/resolution, recovery/resolution with consequences, death, unknown).
Percentage of patients with clinically significant abnormal laboratory tests | On 1 and 14 days of treatment
  Percentage of patients with clinically significant abnormal laboratory tests. Measure is based on the Hematology, blood chemistry, and urinalysis parameters, which are beyond the reference values at the end of treatment.
Changes in Vital Signs (Heart Rate) | On Visit 1 (day 1), Visit 2 (day 4) and Visit 3 (day 8)
  Pulse Rate measured in beats per minute. Based on medical records.
Changes in Vital Signs (Breathing Rate) | On Visit 1 (day 1), Visit 2 (day 4) and Visit 3 (day 8)
  Respiratory Rate measured in breaths per minute. Based on medical records.
Changes in Vital Signs (Axillary temperature) | On Visit 1 (day 1), Visit 2 (day 4) and Visit 3 (day 8)
  Temperature is measured in the armpit using a classic mercury-free thermometer. Based on medical records.

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Gatchina Clinical Interdistrict Hospital, Gatchina
  - Llc "Medlight", Kazan'
  - Specialized Clinical Infectious Diseases Hospital, Krasnodar
  - First Moscow State Medical University named after I.M. Sechenov, Moscow
  - Llc "Diagnosis and Vaccines", Moscow
  - City Children's Clinical Polyclinic # 5, Perm
  - LLC "Professor's Clinic", Perm
  - Clinical and diagnostic center "Health" in Rostov-on-Don, Rostov-on-Don
  - Children's City Polyclinic # 44, Saint Petersburg
  - Children's City Polyclinic # 35, Saint Petersburg
  - Samara Regional Children's Clinical Hospital named after N.N. Ivanova, Samara
  - Saratov City Children's Clinical Hospital, Saratov
  - Clinical Hospital # 2, Yaroslavl
  - Children's City Clinical Hospital # 11, Yekaterinburg